CLINICAL TRIAL: NCT02746042
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial to Assess Efficacy and Safety of the Herbal Medicinal Product Sinupret Extract Coated Tablets in Patients With Chronic Rhinosinusitis
Brief Title: Sinupret Extract Coated Tablets in Chronic Rhinosinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRS-03; 2015-001952-31 (EudraCT Number)
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2017-12

CONDITIONS: Chronic Rhinosinusitis
Keywords: chronic rhinosinusitis; Sinupret extract; herbal medicinal product
MeSH Terms: interventions — Sinupret

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sinupret extract coated tablets (Experimental): Sinupret extract coated tablets: one tablet three times a day orally during the 16-week treatment phase.
  There will be no dose change during the trial.
  Interventions: Drug: Sinupret extract coated tablets
- Placebo coated tablets (Placebo Comparator): Placebo coated tablets: One tablet three times a day orally during the 16-week treatment Phase.
  Interventions: Drug: Placebo coated tablets

INTERVENTIONS:
Drug: Sinupret extract coated tablets — 1 coated tablet 3 times a day for 16-weeks (1-1-1)
  Other Names: Sinupret extract
  Arms: Sinupret extract coated tablets
Drug: Placebo coated tablets — 1 coated tablet 3 times a day for 16-weeks (1-1-1)
  Other Names: Placebo
  Arms: Placebo coated tablets

SUMMARY:
To assess the efficacy of the herbal medicinal product Sinupret extract versus placebo in the treatment of chronic rhinosinusitis (CRS) in adults.

DETAILED DESCRIPTION:
The aim of the present double-blind, placebo-controlled, parallel-group, randomized, phase III clinical trial is to assess the efficacy, safety, and tolerability of Sinupret extract (3 x 160 mg = 480 mg daily) taken for up to 16-weeks compared with placebo in the treatment of chronic rhinosinusitis (CRS) in adults. In addition, in an exploratory approach to identify potential pharmacological modes of action underlying the expected treatment benefit, the anti-inflammatory activity of Sinupret extract will be assessed in a subset of CRS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (IC) including data protection declaration
2. Male and female outpatients aged ≥18 and ≤75 years

   Women will be considered for inclusion if they are not pregnant (as confirmed by urine pregnancy test at V1 and V2), not breastfeeding, or if they are surgically sterile (have had a documented bilateral oophorectomy and/or hysterectomy) or if menopause is ensured (at least 12 months without menstrual bleeding). Women of childbearing potential must use a highly effective (failure rate less than 1% per year, i.e. Pearl Index <1) method of contraception 2 weeks prior to trial inclusion and during the screening/treatment period of the clinical trial (e.g. vasectomized partner, sexual abstinence - the lifestyle of the female has to be such that there is complete abstinence from intercourse from 2 weeks prior to the first dose of trial medication until at least 72 hours after treatment - implants, injectables, combined oral contraceptives, or hormonal intrauterine devices).
3. Diagnosis of bilateral CRS without nasal polyps confirmed by:

   * Nasal endoscopy during the screening phase to confirm inflammation, mucopurulent discharge, and/or edema/mucosal obstruction primarily in middle meatus without nasal polyps being present
   * At the discretion of the investigator, results from a historic imaging diagnostic, i.e. computer tomography (CT), digital volume tomography (DVT), or magnetic resonance tomography (MRT) (before screening and not older than 24 months, not taken during acute exacerbation), which will be considered additionally for confirmation of bilateral involvement of middle meatus and paranasal sinuses without resolution of symptoms (mucosal changes within the ostiomeatal complex and/or sinuses)
4. Bilateral CRS characterized by:

   * Presence of CRS symptoms for >52 weeks prior to enrolment (V1) as documented in the medical file of the patient
   * Major Symptom Score (MSS) ≥10 at V1 and V2 as assessed by the investigator (MSS INV), and rhinorrhea (anterior or posterior) and pain (facial pain or headache) each of at least moderate intensity (score ≥2)

Exclusion Criteria:

1. Sinus surgery within the last 2 years (solitary sinus puncture is allowed)
2. Inferior turbinate reduction (by surgery or other methods) within the last 3 months
3. Presence or history of uni- or bilateral nasal polyps
4. Moderate to severe co-morbid asthma, including allergic asthma
5. Cystic fibrosis
6. Perennial (e.g. patients with clinical symptoms of allergic rhinitis against house dust/mite antigen) or seasonal allergic rhinitis
7. Rhinitis medicamentosa (drug induced rhinitis)
8. Aspirin-exacerbated respiratory disease (aspirin sensitivity)
9. Dentogenic sinusitis or otherwise unilateral sinusitis
10. Presence of anatomical deviations of the nasal septum that significantly impair nasal and paranasal ventilation/airflow
11. Known hypersensitivity to trial medication or excipients
12. Rare hereditary problems of fructose intolerance, galactose intolerance, lactase deficiency, glucose-galactose malabsorption, or sucrase- isomaltase insufficiency
13. Signs or symptoms of acute bacterial sinusitis (e.g. fever >38.5°C, orbital complications, severe unilateral frontal headache, or toothache)
14. Treatment with antihistamines within 4 weeks prior to V1
15. Treatment with 2-3.5% hypertonic saline solution within 2 weeks prior to V1
16. Treatment with systemic or nasal antibiotics or corticosteroids within 4 weeks prior to V1
17. Treatment with decongestant preparations (α-sympathomimetics), analgesics (including systemic non-steroidal inflammatory drugs [NSAIDs], including paracetamol), mucolytics/secretolytics, or alternative medicine preparations for treatment of common cold-like symptoms or with immunomodulating properties within 7 days prior to V1
18. Peptic ulcer
19. Gastritis
20. Other diseases within 5 years prior to V1 that, in the opinion of the investigator, disqualifies the patient for trial enrolment (e.g. liver or kidney disease, severe somatopathic, neurological and/or psychiatric diseases, history of malignancy, alcohol or drug abuse, or immunodeficiency)
21. Parallel participation in another clinical trial, participation in a different trial within less than 6 weeks prior to trial entry, or previous randomization into this clinical trial
22. Known to be, or suspected of being unable to comply with the clinical trial protocol (CTP) that in the opinion of the investigator disqualifies the patient for trial enrolment (e.g. no permanent address, known to be non-compliant, or presenting an unstable psychiatric history)
23. Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope, and possible impact of the clinical trial
24. Patients in custody by juridical or official order
25. Patients who have difficulties in understanding the local language in which the patient information (PI) is given
26. Patients who are members of the staff of the investigational site, staff of the sponsor or involved CRO, the investigator him/herself or close relatives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
MSS-INV at V7 | 16 weeks
  Major Symptom Score (MSS) assessed by the investigator at Visit 7 with Baseline as Covariate; The MSS considers: rhinorrhea [anterior], rhinorrhea [posterior], nasal congestion, headache, and facial pain/pressure

SECONDARY OUTCOMES:
MSS-INV at V4-6 | 12 weeks
  Major Symptom Score (MSS) assessed by the investigator at Visits 4, 5, and 6 with Baseline as Covariate
MSS-PAT at V4-7 | 16 weeks
  Major Symptom Score (MSS) assessed by the Patient at Visits 4, 5, 6, and 7 with Baseline as Covariate
Minimal MSS-INV at V4-7 | 16 weeks
  Minimal Major Symptom Score (MSS) assessed by the Investigator of all visits from Visits 4, 5, 6, and 7
Minimal MSS-PAT at V4-7 | 16 weeks
  Minimal Major Symptom Score (MSS) assessed by the Patient of all visits from Visits 4, 5, 6, and 7
Investigator's Ratings of CRS symptom | 16 weeks
  Investigator's ratings of each individual CRS symptom (i.e. rhinorrhea [anterior], rhinorrhea [posterior], nasal congestion, headache, and facial pain/pressure) at V4, V5, V6, and V7
Patient's Ratings of CRS symptom | 16 weeks
  Patient's ratings of each individual CRS symptom (i.e. rhinorrhea [anterior], rhinorrhea [posterior], nasal congestion, headache, and facial pain/pressure) at V4, V5, V6, and V7
SNOT-22 | 16 weeks
  22-Item Sino-Nasal Outcome Test (SNOT-22)Total Score as well as SNOT-22 primary nasal score (SNOT-22 PNS) and SNOT-22 general quality of life score (SNOT-22 ALQ) at V4, V5, V6, and V7
VAS | 16 weeks
  Total symptom severity assessed by the patient on a visual analogue scale (VAS) at V4, V5, V6, and V7
Responder Rate | 16 weeks
  Proportion of patients whose MSS-INV and MSS-PAT improved by ≥30%, ≥40%, ≥50%, ≥60% and ≥70% at V4, V5, V6, and V7. Responders are defined as patients who show at least an MSS improvement of ≥30%
Concomitant drug and non-drug therapy | 22 weeks
  Patients with permitted concomitant drug and non-drug therapy (i.e. isotonic saline solution as nasal spray, nasal irrigation [nasal lavage], or ultrasonic nebulizer) for CRS
Premature Terminations | 20 weeks
  Number of patients with premature termination due to exacerbation of CRS symptoms
Investigator's and patient's overall assessment of efficacy (questionnaire) | 16 weeks
  At each on-site visit during the treatment phase (V4 to V7), both the investigator and the patient have to provide an overall assessment of treatment efficacy using 5 categories ("very good", "good", "moderate", "poor", and "very poor"; ranges from 0 to 4).
WPAI:GH questionnaire | 22 weeks
  Pharmacoeconomic evaluation (utilization of health care resources) based on "Work Productivity and Activity Impairment, Global Health" (WPAI:GH) questionnaire completed by the patient at V4, V5, V6, and V7
Inflammatory Parameter IL-1beta (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of interleukin-1β (IL-1beta) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter IL-2 (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of interleukin-2 (IL-2) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter IL-4 (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of interleukin-4 (IL-4) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter IL-6 (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of interleukin-6 (IL-6) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter IL-8 (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of interleukin-8 (IL-8) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter IFN-gamma (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of interferon gamma (IFN-gamma) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter TNF-alpha (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of tumor necrosis factor alpha (TNF-alpha) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter MPO (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of myeloperoxidase (MPO) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter ECP (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of eosinophil cationic protein (ECP) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter alpha-2-macroglobulin (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of α2-macroglobulin (alpha-2-macroglobulin) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter HMGB-1 (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of high-mobility group box protein 1 (HMGB-1) in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany
Inflammatory Parameter albumin (nasal secretions: substudy) | 16 weeks
  Absolute concentrations and total amount per sample of albumin in nasal secretions collected at V2, V5, and V7 for a subset of approximately 60 patients in selected investigational sites in Germany

OTHER OUTCOMES:
Safety Endpoints | 22 weeks
  The safety endpoints include:
  1. AEs, SAEs, and treatment-emergent adverse events (TEAEs).
  2. Incidence of adverse drug reactions (ADRs).
  3. Investigator's and patient's overall assessment of tolerability at V7.
  4. Change from baseline (V2) in vital signs after 16 weeks of treatment (V7).
  5. Individual changes from baseline (V2) in safety laboratory parameters after 16 weeks of treatment (V7).
  6. Change from screening (V1) in physical examination (including weight) after 16 weeks of treatment (V7).

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Palm, Dr., Principal Investigator — Praxis Dr. Jürgen Palm, 90552 Röthenbach/Pegnitz, Germany
Locations (36):
- Germany (18):
  - Bionorica Investigative Site, Berlin
  - Bionorica Investigative Site, Braunschweig
  - Bionorica Investigative Site, Chemnitz
  - Bionorica Investigative Site, Dresden
  - Bionorica Investigative Site, Duisburg
  - Bionorica Investigative Site, Essen
  - Bionorica Investigative Site, Frankfurt am Main
  - Bionorica Investigative Site, Göttingen
  - Bionorica Investigative Site, Heidelberg
  - Bionorica Investigative Site, Markkleeberg
  - Bionorica Investigative Site, Mittweida
  - Bionorica Investigative Site, Munich
  - Bionorica Investigative Site, Neuenhagen
  - Bionorica Investigative Site, Nuremberg
  - Bionorica Investigative Site, Röthenbach/Pegnitz
  - Bionorica Investigative Site, Schlüchtern
  - Bionorica Investigative Site, Schorndorf
  - Bionorica Investigative Site, Wuppertal
- Poland (18):
  - Bionorica Investigative Site, Bialystok
  - Bionorica Investigative Site, Bydgoszcz
  - Bionorica Investigative Site, Gdansk
  - Bionorica Investigative Site, Gdynia
  - Bionorica Investigative Site, Katowice
  - Bionorica Investigative Site, Kielce
  - Bionorica Investigative Site, Krakow
  - Bionorica Investigative Site, Limanowa
  - Bionorica Investigative Site, Lodz
  - Bionorica Investigative Site, Lublin
  - Bionorica Investigative Site, Piaseczno
  - Bionorica Investigative Site, Szczecin
  - Bionorica Investigative Site, Tychy
  - Bionorica Investigative Site, Warsaw
  - Bionorica Investigative Site, Wieliczka
  - Bionorica Investigative Site, Wroclaw
  - Bionorica Investigative Site 222, Zgierz
  - Bionorica Investigative Site 224, Zgierz

IPD SHARING:
Plan to Share IPD: No
It is currently not planned to annex individual participant data (IPD) to publications of the study results.